CLINICAL TRIAL: NCT06981000
Title: A Feasibility Study of Locally Adapted Nature-based Health Interventions for People With Mild to Moderate Anxiety, Depression and Stress
Brief Title: A Feasibility Study of Nature-based Health Interventions for People With Mild to Moderate Anxiety, Depression and Stress
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Collaborators: DEFACTUM, Central Denmark Region, Denmark (Unknown); Department of Public Health, Aarhus University, Denmark (Unknown); Research Unit for General Practice, Aarhus, Denmark (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 514-0614/25-5000
Record Dates: First submitted 2025-03-14; First posted 2025-05-20 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Anxiety; Anxiety Disorders; Depression - Major Depressive Disorder; Depressive Disorder; Stress, Psychologic
Keywords: Nature-based health intervention; Mental health; Anxiety; Depression; Stress-related disorders
MeSH Terms: conditions — Anxiety Disorders; Depressive Disorder; Stress, Psychological; Psychological Well-Being; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Nature-based health intervention (Other): This is a single-arm feasibility study of locally adapted NBHIs
  Interventions: Behavioral: Locally adapted nature-based health intervention

INTERVENTIONS:
Behavioral: Locally adapted nature-based health intervention — The locally adapted NBHIs are organized according to the following structure:
  * Duration of the program: Minimum 10 weeks, once a week, 1.5-2.5 hours per session
  * Group composition: Across conditions: mild to moderate anxiety, depression, and/or stress
  * Group size: 8-12 participants in a closed group
  In the locally adapted programs, activities in nature are based on three main mechanisms of change (nature interaction and sensory experiences, social communities, and physical activity and movement).

SUMMARY:
Background and aimThe increased burden on mental health both globally and nationally is a serious challenge that requires attention and action from healthcare professionals, politicians, and decision-makers. According to the report "The National Health Profile 2021" from the Danish Health Authority, the number of adult Danes (over 16 years) with a low mental health score has increased by seven percentage points from 2010-2021 and now stands at 17.4%. A significant proportion of these individuals suffer from anxiety, depression, and/or stress. This increase in people with reduced mental health has consequences both for the individual's quality of life and for society as a whole. Thus, more than 13% of the Danish population is prescribed medication for the treatment of mental illnesses, and only 28% of them are able to work while experiencing their illness.There is a growing recognition that the challenges associated with mental health cannot be solved solely through clinical treatment or medication. In order to offer citizens and patients the best possible support, it is important to look for sustainable solutions to promote mental health and ensure access to effective treatment options. Despite a significant increase in the number of published research studies on the positive impact of nature on mental health, there has not previously been developed a theoretical foundation and a comprehensive evidence base for nature-based health interventions in a Danish context, and there has been a lack of a structured and systematically developed understanding of the mechanisms of change in nature-based health interventions (NBHIs), so they can be implemented in a way that aligns with the best available knowledge in the field.In phase 1 of the project, a systematic review of the literature has been conducted. Hereby followed an extensive co-creation process, including the development of a logic model and an underlying program theory, and established collaboration with three relevant implementation partners.In phase 2 of the project, the aim was to test the feasibility of three locally adapted NBHIs in a feasibility study with up to 120 participants (40 participants per partner) at three different partners. MethodsThe locally adapted NBHIs will be tested at the Psychiatric Center Glostrup and at the Kolding and Silkeborg municipal health centers from March to November 2025. The intervention will be carried out as an interdisciplinary initiative facilitated by two healthcare professionals employed at the respective partners, who already have experience in delivering NBHIs to the target group.The NBHIs are organized according to the following structure:• Duration of the program: Minimum 10 weeks, once a week, 1.5-2.5 hours per session• Group composition: Across conditions: mild to moderate anxiety, depression, and/or stress• Group size: 8-12 participants in a closed groupIn the locally adapted programs, activities in nature are based on three main mechanisms of change (nature interaction and sensory experiences, social communities, and physical activity and movement), identified in phase 1 of the project. The healthcare professionals responsible for the programs will tailor the activities individually. All activities are designed based on a generic logic model, developed through a co-creation process.Safety plays a central role in the nature-based health interventions. All activities are planned with a focus on the participants' physical and mental well-being. Potential risks are assessed and minimized through the selection of suitable natural environments, appropriate equipment, and thorough instruction. The healthcare professionals ensure a safe environment where participants can feel comfortable, both physically and psychologically. Additionally, accessibility and any individual needs are considered, so all participants can safely engage in the activities. With this study, the results of a new treatment or examination will not be conduced (and none of the participants will receive a worse treatment offer than what currently exists). It is about investigating the feasibility of locally adapted NBHIs at three different partners who already have nature-based programs.Both quantitative and qualitative data will be collected. These will include questionnaire data, data from registration of participation by the partner, participant observation, focus group interviews with participants from the NBHIs, as well as focus group interviews with the healthcare professionals who are carrying out the NBHIs. As part of the qualitative research, experiences with and perceptions of the process, including the feasibility of the NBHI and how the participants respond to the intervention will be examended. Written consent will be obtained from the participants and healthcare professionals prior to this.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or above
* Diagnosed with or symptoms of mild to moderate anxiety, depression, and/or experiencing symptoms of stress, and as a result is the primary cause of reduced functionality
* Contact through health center in the municipality, general practitioner, job center, self-referral, or via outpatient psychiatric rehabilitation plan
* Sick leave is not a requirement

Exclusion Criteria:

* Age less than 18 years
* Serious psychiatric disorders like schizophrenia, bipolar disorder, severe anxiety or depression, posttraumatic stress disorder (PTSD)
* Suicidal risk
* Alcohol or substance abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2025-11-24 (Estimated); Study Completion 2025-11-24 (Estimated)

PRIMARY OUTCOMES:
Ability to enroll participants who meet the inclusion criteria within the target time frame | From enrollment to the end of the treatment at 10 weeks
  Number of participants recruited
Population composition | From enrollment to the end of the treatment at 10 weeks
  The composition of participants with symptoms of anxiety, depression and stress, respectively, reported in the questionnaire data
Non-participation | From enrollment to the end of the treatment at 10 weeks
  Registration by the health care team of reasons for declining to participate in the nature-based health intervention
Participant adherence to the intervention | From enrollment to the end of the treatment at 10 weeks
  How many times out of 10 sessions do the participants participate, reported in the questionnaire data
Which adaptions are conducted during the program | From enrollment to the end of the treatment at 10 weeks
  Registrations by the health care team
Which components from the generic logic model come into play | From enrollment to the end of the treatment at 10 weeks
  Qualitatively data through participant observation and focus group interviews with the health care team
Are the right mechanisms of change from the logic model identified and incorporated in the intervention | From enrollment to the end of the treatment at 10 weeks
  Qualitatively data through participant observation and focus group interviews with the health care team
What was the participants' perception of the intervention? | Week 11, one week after the completion of the intervention
  Qualitatively data through focus group interviews with the participants
What was the health care teams' perception of the intervention? | From enrollment to the end of the treatment at 10 weeks
  Qualitatively data through focus group interviews with the health care team

SECONDARY OUTCOMES:
Mental well-being | Baseline, post program (after 10 weeks)
  WHO-5 Well-being Index. Five item scale answered on a Likert scale 0-5, with a lower score indicating worse outcome
Symptoms of anxiety, depression and/or stress | Baseline, post program (after 10 weeks)
  Depression, Anxiety and Stress Scale (DASS-21). 21 item scale answered on a Likert scale 0-3, with a higher score indicating worse outcome
Life quality | Baseline, post program (after 10 weeks)
  Satisfaction with Life Scale. Five item scale answered on a Likert scale 1-7, with a lower score indicating worse outcome
Nature relatedness | Baseline, post program (after 10 weeks)
  Environmental Identity Scale. 14 item scale answered on a Likert scale 1-7, with a lower score indicating lower nature relatedness

CONTACTS AND LOCATIONS:
Overall Officials: Dorthe V Poulsen, Ass professor, Study Director — Department of Geosciences and Natural Resource Management, University of Copenhagen, Denmark
Locations (1):
- Department of Geosciences and Natural Resource Management, University of Copenhagen, Denmark, Copenhagen, Denmark, Denmark

IPD SHARING:
Plan to Share IPD: No